CLINICAL TRIAL: NCT00054652
Title: Survey of Sensory and Motor Tricks in Focal Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030089; 03-N-0089
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-02

CONDITIONS: Focal Dystonia
Keywords: Geste Antagoniste; TMS; Sensorimotor Integration; Writer's Cramp; Sensory Input; Focal Dystonia
MeSH Terms: conditions — Dystonic Disorders

SUMMARY:
This study will collect information on (tricks) patients with focal dystonia use to relieve their symptoms. Dystonia is a movement disorder caused by sustained muscle contractions often causing twisting and abnormal posturing. Dystonia may be generalized, affecting at least one leg and the trunk of the body, segmental, affecting adjacent body parts, or focal, affecting a single body part, such as the hand or eyelid. It may be task-specific, such as writer's, musician's or sportsman's cramps. Some patients with focal dystonia use (tricks), such as touching the face or hand, to stop or alleviate the abnormal movement. This study will survey the types of tricks people with focal dystonia use in order to learn more about the disorder.

Patients 18 years of age and older with focal dystonia may be eligible for this study. Candidates will be screened for eligibility with a medical history, clinical evaluation, and review of their medical records.

In one 30- to 45-minute clinic visit, participants will be interviewed about their dystonia symptoms and the tricks they use to relieve the symptoms. They may be asked to show the investigators how the tricks work

DETAILED DESCRIPTION:
The purpose of this study is to collect and organize information concerning a phenomenon known as 'sensory tricks' or Geste antagoniste in focal dystonia. Sensory tricks, which we will refer to as 'tricks' since some involve motor as well as sensory input, are various stimuli used by dystonic patients to transiently diminish their spasms (Jankovic and Fahn 1993). The phenomenon of tricks is evidence for the abnormality of sensorimotor integration in focal dystonia, yet it is little studied or understood. A survey of the history and characteristics of tricks will lead to a better understanding of this puzzling phenomenon, and a step toward the understanding of the mechanism of focal dystonia.

ELIGIBILITY:
INCLUSION CRITERIA

Patients with focal dystonia diagnosed by review of medical record, history, and clinical evaluation.

EXCLUSION CRITERIA

Any individual without focal dystonia.

Any individual who is unable to provide accurate history, or is critically ill.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2003-02; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States